CLINICAL TRIAL: NCT01052532
Title: The Study to Define the Unique Molecular Mechanisms of Mitral Regurgitation in Order to Find New Targeted Therapy to Attenuate the Remodeling and Delay the Need for Surgery and Improve Surgical Outcomes.
Brief Title: Molecular Mechanisms of Mitral Regurgitation-Aim 2
Acronym: P1A2
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Louis J. Dell'Italia, MD, UAB
Other Study IDs: F0400105007
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Mitral Regurgitation
Keywords: Mitral Regurgitation; LV remodeling; Reactive nitrogen species; Cardiac MRI; Adrenergic overdrive
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, myocyte tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitral Regurgitation pre&post operation: Patients with severe Mitral Regurgitation without evidence of ischemia are tested prior to surgery and after valve repair.

SUMMARY:
The investigators hypothesize that MR in humans is characterized by adrenergic overdrive, reactive nitrogen species, and an antifibrotic phenotype that relate to the severity of adverse LV remodeling prior to surgery and outcome after valve repair.

DETAILED DESCRIPTION:
In Western society, the most common causes of chronic nonischemic mitral regurgitation (MR) is myxomatous degeneration of the valve.Unlike pressure overload, where fibrosis reduction and renin-angiotensin system (RAS) blockade is beneficial, the dynamics of extracellular matrix homeostasis in volume overload produce minimal changes in collagen content. It is for this reason that RAS blockade is not beneficial in patients and in animal models with pure volume overload of MR. In particular, we have shown that ACE inhibition, which increases cardiac interstitial bradykinin-resulting in a reduction in collagen production and activation of matrix metalloproteinase (MMP)-is particularly harmful in volume overload. Further, we showed that MR in the dog is marked by an early and persistent decrease in LV interstitial collagen and MMP activation, as well as the expression of bradykinin. Thus, therapies targeted at matrix reduction may exacerbate the disease process by decreasing the collagen connections between cardiomyocytes.

Another important pathophysiologic mechanism in the adverse LV remodeling in MR is the adrenergic nervous system and inflammation. It is of interest that we and others have found increased adrenergic drive to be an important early mechanism in the volume overload of MR in dogs and MR in patients. This response can be attributed to the early recruitment of preload reserve in adaptation to the volume load. In fact, beta1-adrenergic receptor (AR) blockade improved LV remodeling, attenuated matrix degradation, and improved LV and cardiomyocyte function in the dog with MR. Increased adrenergic stimulation can also lead to the generation of reactive nitrogen species and TNF-alpha that, in turn, can activate MMPs, thereby perpetuating the cycle of matrix degradation and adverse LV remodeling.

The investigators hypothesize that MR in humans is characterized by adrenergic overdrive, reactive nitrogen species, and an antifibrotic phenotype that relate to the severity of adverse LV remodeling prior to surgery and outcome after valve repair.

Aim 1. To show that regional stress and strain of MR relates to indices of adrenergic efferent innervation and function of the LV myocardium. LV tissue will be analyzed for innervation density, catecholamine content and reuptake, and beta1- and beta2-AR density.

Aim 2. To define the extent and nature of reactive nitrogen species production in LV myocardium and determine whether peripheral plasma measurements correlate with myocardial origin. LV tissue and plasma will be analyzed for the extent of protein thiol oxidation and protein tyrosine nitration and myeloperoxidase and xanthine oxidase activities.

Aim 3. To show increased expression of antifibrotic factors in LV myocardium and that peripheral plasma measurements correlate with myocardial origin and whether these factors correlate with functional recovery by MRI. LV tissue will be analyzed for MT1MMP, MMP-1,-2 and -9, bradykinin type-2 receptor, AT1 and AT2 receptor, collagen type II and III and plasma will be analyzed for collagen breakdown products.

Currently, there is no recommended therapy for the pure volume overload of mitral regurgitation, these studies will define the unique molecular mechanisms that will lead to new targeted therapy to attenuate the remodeling and delay the need for surgery and improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old or older.
2. Severe MR by echo or catheterization without evidence of ischemia requiring surgery documented by cardiac catheterization and/or maximal stress test with myocardial perfusion imaging.

Exclusion Criteria:

1. Significant obstructive coronary artery disease and/or myocardial ischemia on graded exercise test with myocardial perfusion.
2. Previous myocardial infarction.
3. Hypertrophic cardiomyopathy, congenital or pericardial disease.
4. Aortic valve disease (> trace aortic regurgitation or mean gradient > 10 mmHg)
5. Mitral stenosis (mean gradient > 5 mmHg, valve area < 1.5 cm2).
6. Renal failure with creatinine > 2.5 mg/dl.
7. Renal artery stenosis.
8. Severe comorbidity such as liver disease, malignancy, collagen vascular disease, or chronic steroid requirement.
9. Pregnancy (negative pregnancy test and effective contraceptive methods are required prior to enrollment of females of childbearing potential (not post-menopausal or surgically sterilized).

Exclusion Criteria Related to MRI

1. Severe claustrophobia.
2. Presence of a pacemaker or non-removable hearing aid.
3. Presence of metal clips in the body.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ptaients scheduled for Mitral valve repair from c ardiology clinic / Hospital
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2005-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma levels of MT1MMP, MMP-1,-2 and -9, bradykinin type-2 receptor, AT1 and AT2 receptor, collagen type II and III and collagen breakdown products | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis J Dell'Italia, M.D, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] 1. Dell'Italia LJ. Mitral Regurgitation. In Hurst The Heart. Eds. O'Rourke, Sclhant, Alexader, Fuster. 11th Edition, Chapter 57 pp 1169-1695, 2004.
- [Background] Olson LJ, Subramanian R, Ackermann DM, Orszulak TA, Edwards WD. Surgical pathology of the mitral valve: a study of 712 cases spanning 21 years. Mayo Clin Proc. 1987 Jan;62(1):22-34. doi: 10.1016/s0025-6196(12)61522-5. PMID 3796056
- [Background] Borer JS, Bonow RO. Contemporary approach to aortic and mitral regurgitation. Circulation. 2003 Nov 18;108(20):2432-8. doi: 10.1161/01.CIR.0000096400.00562.A3. No abstract available. PMID 14623790
- [Background] Wisenbaugh T, Essop R, Rothlisberger C, Sareli P. Effects of a single oral dose of captopril on left ventricular performance in severe mitral regurgitation. Am J Cardiol. 1992 Feb 1;69(4):348-53. doi: 10.1016/0002-9149(92)90232-n. PMID 1734647
- [Background] Rothlisberger C, Sareli P, Wisenbaugh T. Comparison of single dose nifedipine and captopril for chronic severe mitral regurgitation. Am J Cardiol. 1994 May 15;73(13):978-81. doi: 10.1016/0002-9149(94)90148-1. No abstract available. PMID 8184862
- [Background] Wisenbaugh T, Sinovich V, Dullabh A, Sareli P. Six month pilot study of captopril for mildly symptomatic, severe isolated mitral and isolated aortic regurgitation. J Heart Valve Dis. 1994 Mar;3(2):197-204. PMID 8012639
- [Background] Marcotte F, Honos GN, Walling AD, Beauvais D, Blais MJ, Daoust C, Lisbona A, McCans JL. Effect of angiotensin-converting enzyme inhibitor therapy in mitral regurgitation with normal left ventricular function. Can J Cardiol. 1997 May;13(5):479-85. PMID 9179087
- [Background] Host U, Kelbaek H, Hildebrandt P, Skagen K, Aldershvile J. Effect of ramipril on mitral regurgitation secondary to mitral valve prolapse. Am J Cardiol. 1997 Sep 1;80(5):655-8. doi: 10.1016/s0002-9149(97)00445-1. PMID 9295005
- [Background] Tischler MD, Rowan M, LeWinter MM. Effect of enalapril therapy on left ventricular mass and volumes in asymptomatic chronic, severe mitral regurgitation secondary to mitral valve prolapse. Am J Cardiol. 1998 Jul 15;82(2):242-5. doi: 10.1016/s0002-9149(98)00325-7. PMID 9678300
- [Background] Dujardin KS, Enriquez-Sarano M, Bailey KR, Seward JB, Tajik AJ. Effect of losartan on degree of mitral regurgitation quantified by echocardiography. Am J Cardiol. 2001 Mar 1;87(5):570-6. doi: 10.1016/s0002-9149(00)01433-8. PMID 11230841
- [Background] Gaasch WH, Aurigemma GP. Inhibition of the renin-angiotensin system and the left ventricular adaptation to mitral regurgitation. J Am Coll Cardiol. 2002 Apr 17;39(8):1380-3. doi: 10.1016/s0735-1097(02)01766-7. No abstract available. PMID 11955859
- [Background] Stewart JA Jr, Wei CC, Brower GL, Rynders PE, Hankes GH, Dillon AR, Lucchesi PA, Janicki JS, Dell'Italia LJ. Cardiac mast cell- and chymase-mediated matrix metalloproteinase activity and left ventricular remodeling in mitral regurgitation in the dog. J Mol Cell Cardiol. 2003 Mar;35(3):311-9. doi: 10.1016/s0022-2828(03)00013-0. PMID 12676546
- [Background] Nemoto S, Hamawaki M, De Freitas G, Carabello BA. Differential effects of the angiotensin-converting enzyme inhibitor lisinopril versus the beta-adrenergic receptor blocker atenolol on hemodynamics and left ventricular contractile function in experimental mitral regurgitation. J Am Coll Cardiol. 2002 Jul 3;40(1):149-54. doi: 10.1016/s0735-1097(02)01926-5. PMID 12103269
- [Background] Dell'italia LJ, Balcells E, Meng QC, Su X, Schultz D, Bishop SP, Machida N, Straeter-Knowlen IM, Hankes GH, Dillon R, Cartee RE, Oparil S. Volume-overload cardiac hypertrophy is unaffected by ACE inhibitor treatment in dogs. Am J Physiol. 1997 Aug;273(2 Pt 2):H961-70. doi: 10.1152/ajpheart.1997.273.2.H961. PMID 9277516
- [Background] Perry GJ, Wei CC, Hankes GH, Dillon SR, Rynders P, Mukherjee R, Spinale FG, Dell'Italia LJ. Angiotensin II receptor blockade does not improve left ventricular function and remodeling in subacute mitral regurgitation in the dog. J Am Coll Cardiol. 2002 Apr 17;39(8):1374-9. doi: 10.1016/s0735-1097(02)01763-1. PMID 11955858
- [Background] Nagatsu M, Zile MR, Tsutsui H, Schmid PG, DeFreyte G, Cooper G 4th, Carabello BA. Native beta-adrenergic support for left ventricular dysfunction in experimental mitral regurgitation normalizes indexes of pump and contractile function. Circulation. 1994 Feb;89(2):818-26. doi: 10.1161/01.cir.89.2.818. PMID 8313571
- [Background] Tallaj J, Wei CC, Hankes GH, Holland M, Rynders P, Dillon AR, Ardell JL, Armour JA, Lucchesi PA, Dell'Italia LJ. Beta1-adrenergic receptor blockade attenuates angiotensin II-mediated catecholamine release into the cardiac interstitium in mitral regurgitation. Circulation. 2003 Jul 15;108(2):225-30. doi: 10.1161/01.CIR.0000079226.48637.5A. Epub 2003 Jul 7. PMID 12847066
- [Background] Hankes GH, Ardell JL, Tallaj J, Wei CC, Aban I, Holland M, Rynders P, Dillon R, Cardinal R, Hoover DB, Armour JA, Husain A, Dell'Italia LJ. Beta1-adrenoceptor blockade mitigates excessive norepinephrine release into cardiac interstitium in mitral regurgitation in dog. Am J Physiol Heart Circ Physiol. 2006 Jul;291(1):H147-51. doi: 10.1152/ajpheart.00951.2005. PMID 16772522
- [Background] Tsutsui H, Spinale FG, Nagatsu M, Schmid PG, Ishihara K, DeFreyte G, Cooper G 4th, Carabello BA. Effects of chronic beta-adrenergic blockade on the left ventricular and cardiocyte abnormalities of chronic canine mitral regurgitation. J Clin Invest. 1994 Jun;93(6):2639-48. doi: 10.1172/JCI117277. PMID 7911128
- [Background] Mehta RH, Supiano MA, Oral H, Grossman PM, Montgomery DS, Smith MJ, Starling MR. Compared with control subjects, the systemic sympathetic nervous system is activated in patients with mitral regurgitation. Am Heart J. 2003 Jun;145(6):1078-85. doi: 10.1016/S0002-8703(03)00111-X. PMID 12796766
- [Background] Mehta RH, Supiano MA, Oral H, Grossman PM, Petrusha JA, Montgomery DG, Briesmiester KA, Smith MJ, Starling MR. Relation of systemic sympathetic nervous system activation to echocardiographic left ventricular size and performance and its implications in patients with mitral regurgitation. Am J Cardiol. 2000 Dec 1;86(11):1193-7. doi: 10.1016/s0002-9149(00)01201-7. PMID 11090790
- [Background] Oral H, Sivasubramanian N, Dyke DB, Mehta RH, Grossman PM, Briesmiester K, Fay WP, Pagani FD, Bolling SF, Mann DL, Starling MR. Myocardial proinflammatory cytokine expression and left ventricular remodeling in patients with chronic mitral regurgitation. Circulation. 2003 Feb 18;107(6):831-7. doi: 10.1161/01.cir.0000049745.38594.6d. PMID 12591752
- [Background] Siwik DA, Colucci WS. Regulation of matrix metalloproteinases by cytokines and reactive oxygen/nitrogen species in the myocardium. Heart Fail Rev. 2004 Jan;9(1):43-51. doi: 10.1023/B:HREV.0000011393.40674.13. PMID 14739767